CLINICAL TRIAL: NCT05395767
Title: A Prospective Cohort Study of Skeletally Immature Patients Requiring Endoscopic Anterior Cruciate Ligament Reconstruction, Using Living Donor Hamstring Allograft From a Parent
Brief Title: LIVing Donor Allograft for Anterior Cruciate Ligament Reconstruction Study
Acronym: LivD_ACLR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maidstone & Tunbridge Wells NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MaidstoneNHS
Record Dates: First submitted 2021-12-02; First posted 2022-05-27 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-11

CONDITIONS: ACL

STUDY DESIGN:
Intervention Model Description: Cohort Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endoscopic ACL reconstruction with parent allograft tendon (Experimental)
  Interventions: Procedure: Endoscopic Anterior Cruciate Ligament reconstruction using living donor hamstring allograft from a parent donor

INTERVENTIONS:
Procedure: Endoscopic Anterior Cruciate Ligament reconstruction using living donor hamstring allograft from a parent donor — The Parent donor will undergo hamstring tendon graft harvest under general anaesthesia in a routine fashion in one theatre. The Graft material will be transported thorough to the adjacent theatre, where the child will be anaesthetised and undergoing arthroscopy of their injured knee in preparation for receiving the graft. ACL reconstruction Surgery will be undertaken in the child recipient as per the Surgeons usual technique, +/- meniscus repair +/- lateral tenodesis as required.

SUMMARY:
The Anterior Cruciate Ligament (ACL) is a major stabiliser of the knee. ACL rupture is being increasingly identified in children and skeletally immature patients. The current advice in younger patients is usually to undergo ACL reconstruction. The choice of an ideal graft in children is difficult

This study will use a technique involves the use of hamstring tendons from a living donor, where the adult (usually a parent) agrees to donate their hamstring tendons, which are dissected out of them and implanted into the child

DETAILED DESCRIPTION:
The Anterior Cruciate Ligament (ACL) is a major stabiliser of the knee. ACL rupture is being increasingly identified in children and skeletally immature patients. Following rupture of this ligament, the current advice in younger patients is usually to undergo ACL reconstruction. Different tissue or materials can be used to reconstruct the ligament. In the majority of cases around the world, tendon material taken from somewhere else in the patient is preferred, particularly the hamstring or patellar tendons.

The choice of an ideal graft in children is difficult. Patients who have not fully grown have smaller tendons than adults, making them less suitable for use in reconstructive surgery. Another option for children's reconstructions is allograft - tendons taken from another human being. This has most commonly been from organ donation (taking tendons from a recently deceased individual) however the rerupture rate of allograft has been shown to be higher than in autograft (tendons taken from the patient themselves). The higher rate of rerupture may be related to the sterilising and storage processes of the harvested tendons.

This study will use a technique used by a leading hospital in Sydney, Australia, that sees and treats a large volume of these patients and has published good outcomes. The technique involves the use of hamstring tendons from a living donor, where the adult (usually a parent) agrees to donate their hamstring tendons, which are dissected out of them and implanted into the child. The technique has the advantage of leaving the child's own tendons intact, and having a larger sized tendon from a parent.

Patients & parents will be approached in clinic after MRI confirmation of an ACL rupture. If all inclusion and exclusion criteria have been passed and they consent to participate, screening documents & tests will be completed. The parent will undergo a hamstring tenotomy whilst the child is prepped for ACL reconstruction, then the hamstring donor graft will be inserted in the child patient, using the surgeon's routine fixation devices. All patients will be assessed for skeletal maturity prior to surgery and will be followed up for two years or until skeletal maturity, whichever happens latest. They will follow standard rehabilitation guidelines for paediatric patients at Maidstone & Tunbridge Wells National Health Service Trust (MTW NHS Trust) and be seen at set study intervals for clinical review, subjective and objective assessment. Any adverse events will be reported to the health regulation authority and Human Tissue Licence Authority.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8 to 17 years inclusive and have a clinically and radiologically confirmed ACL rupture that requires reconstruction.
* Patients who have had previous surgery for meniscal pathology .
* Patients with current meniscal pathology
* The child and their responsible adult are in agreement with the choice to undergo anterior cruciate ligament reconstruction using living donor allograft.
* Donors has not previously undergone tendon harvest on the chosen donor limb
* Patients are willing to attend follow up appointments and agree to fill in knee questionnaires and allow instrumented knee ligament testing.

Exclusion Criteria:

* Patients who have previously undergone ACL surgery on the same limb (and therefore require revision surgery)
* Patients who are immunosuppressed, or receiving immunosuppressive therapy
* Patients who are unable to attend follow-up appointments for continued research purposes.
* Donors who have previously undergone hamstring tendon surgery on the donor limb
* Patients and donors who have a positive screening blood test for any of the transmissible infections tested
* Donors whose answers to the 'Donor Documentation Questionnaire' indicate that there could be a risk of transmissible infection, may not included
* Donors who are not considered healthy enough to undergo a tenotomy under General anaesthetic

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee Subjective Knee Form (IKDC) | 6 weeks post op
  Evaluates symptoms, daily activity and sports function. Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
International Knee Documentation Committee Subjective Knee Form (IKDC) | 6 months post op
  Evaluates symptoms, daily activity and sports function. Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
International Knee Documentation Committee Subjective Knee Form (IKDC) | 1 year post op
  Evaluates symptoms, daily activity and sports function
International Knee Documentation Committee Subjective Knee Form (IKDC) | 2 years post op
  Evaluates symptoms, daily activity and sports function. Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Tegner Lysholm | 6 weeks post op
  Symptom reporting questionnaire made up of two components. The Lysholm score Scores range from 0 (worse disability) to 100 (less disability) and the Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Lysholm | 6 months post op
  Symptom reporting questionnaire made up of two components. The Lysholm score Scores range from 0 (worse disability) to 100 (less disability) and the Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Lysholm | 1 year post op
  Symptom reporting questionnaire made up of two components. The Lysholm score Scores range from 0 (worse disability) to 100 (less disability) and the Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Lysholm | 2 years post op
  Symptom reporting questionnaire made up of two components. The Lysholm score Scores range from 0 (worse disability) to 100 (less disability) and the Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.

SECONDARY OUTCOMES:
KT 1000 | 1 year post op
  instrumented laxity test
KT 1000 | 2 years post op
  instrumented laxity test
return to sport questionnaire | 1 year post op
  Psychological readiness for return to sport questionnaire, comprises 12 questions with a score of 1 to 10 for each. Where a lower score means a better outcome.
return to sport questionnaire | 2 years post op
  Psychological readiness for return to sport questionnaire, comprises 12 questions with a score of 1 to 10 for each. Where a lower score means a better outcome.
hop test | 1 year post op
  functional test, In this test, the aim is to jump as far as possible on a single leg, without losing balance and landing firmly. The distance is measured from the start line to the heel of the landing leg. The goal is to have a less than 10% difference in hop distance between the injured limb and uninjured limb.
hop test | 2 years post op
  functional test, In this test, the aim is to jump as far as possible on a single leg, without losing balance and landing firmly. The distance is measured from the start line to the heel of the landing leg. The goal is to have a less than 10% difference in hop distance between the injured limb and uninjured limb.
squat test | 6 months post op
  functional test, scoring of the movement strategy occurring in individual body regions, where 0 for appropriate strategy and one for inappropriate movements, for each region with best overall score being 0 and worst 10 points
squat test | 1 year post op
  functional test, scoring of the movement strategy occurring in individual body regions, where 0 for appropriate strategy and one for inappropriate movements, for each region with best overall score being 0 and worst 10 points
squat test | 2 years post op
  functional test, scoring of the movement strategy occurring in individual body regions, where 0 for appropriate strategy and one for inappropriate movements, for each region with best overall score being 0 and worst 10 points

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Bowman, Principal Investigator — Maidstone & Tunbridge Wells NHS Trust
Locations (1):
- Trauma & Orthopaedic Dept, Tunbridge Wells Hospital, Pembury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No